CLINICAL TRIAL: NCT03384290
Title: A Dose Escalating Single Blind Study to Assess the Safety, Tolerability and Pharmacokinetics of a Single Dose of PRS-060 Administered by Oral Inhalation or IV Infusion in Healthy Subjects
Brief Title: Study of a Single Dose of PRS-060 Administered by Oral Inhalation or IV Infusion in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pieris Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRS-060-PCS_06_17
Record Dates: First submitted 2017-11-26; First posted 2017-12-27 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Healthy Subjects
Keywords: Asthma; Anticalin; PRS-060; Healthy Volunteers; Pieris; IL-4 receptor alpha; IL-13; IL-4
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Single Group Assignment This is a phase 1, dose escalating study to assess safety, tolerability, and PK of a single dose of PRS-060 administered by oral inhalation or IV infusion to healthy male and female subjects. This study will be conducted utilizing a single-blind, randomized, dose-escalating design.
Who Masked: Participant
Masking Description: Randomization is assigned by the pharmacist according to predetermined randomization code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PRS-060 (Experimental)
  Interventions: Drug: PRS-060

INTERVENTIONS:
Drug: PRS-060 — Drug
  Arms: PRS-060
Drug: Placebo — PRS-060 Matching Placebo
  Arms: Placebo

SUMMARY:
A Dose Escalating Study of PRS-060 Administered by Oral Inhalation or IV Infusion in Healthy Subjects

DETAILED DESCRIPTION:
PRS-060 is a new drug being developed for treatment of asthma. The main purpose of this study is to investigate the safety, tolerability and pharmacokinetics of single ascending doses of PRS-060 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female of non-childbearing potential (post-menopausal or surgically sterilized) subjects of 18 to 55 years of age
* Body mass index (BMI) of 18-35
* Subjects who are non-smokers or ex-smokers who have not smoked in the last 6 months (determined by urine cotinine < 500 ng/ml, at screening visit).

Exclusion Criteria:

* History or clinical manifestations of any clinically significant medical disorder that, in the opinion of the investigator, may put the subject at risk because of participation in the study, influence the results of the study or affect the subject's ability to participate in the study.
* A history of drug or alcohol abuse.
* History of, or known significant infection including hepatitis A, B, or C, Human immunodeficiency Virus (HIV), tuberculosis (i.e., positive result for Interferon (INF)-y release assay (IGRA), QuantiFERON TB-Gold), that may put the subject at risk during participation in the study.
* Any clinically significant illness, infection, medical/surgical procedure, or trauma within 4 weeks of day 1 or planned inpatient surgery or hospitalization during the study period.
* Subjects with any history of malignancy or neoplastic disease.
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, as judged by the principal investigator.
* Subjects who have received live or attenuated vaccine in the 4 weeks prior to day 1 subjects with a disease history suggesting abnormal immune function
* Inability to communicate well with the Investigator (i.e. language problem, poor mental development or impaired cerebral function)
* Participation in any clinical study for a New Chemical Entity within the previous 16 weeks or a marketed drug clinical study within the previous 12 weeks or within 5 half- lives, whichever is the longer, before the first dose of study drug.
* Donation of 450 ml or more blood within the previous 12 weeks
* Women who are pregnant
* Males who are sexually active with a female partner of childbearing potential and who have not had a vasectomy and who do not agree to double methods of contraception with at least one barrier from day 1 for 90 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) after a single inhaled or IV infusion dose of PRS-060. | From time of dose until 30 days after dosing.
  The number of participants with treatment related AEs as assessed by CTCAE v4.0. Subjects will be monitored for AEs during study participation (beginning at the time study drug is first administered) until 30 days after dosing.
Change in blood pressure. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess blood pressure (systolic and diastolic) as a criterion of safety and tolerability variables.
Change in heart rate. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in beats per minute (BPM) as a criterion of safety and tolerability variables.
Change in body temperature. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in body temperature as a criterion of safety and tolerability variables as measure in degrees Celsius.
Change in electrocardiograms (ECGs). | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in cardiovascular system function (change in QTC parameters) as a criterion of safety and tolerability variables.
Change in FEV1 (Forced expiratory volume 1-second) | Pre-dose and post-dose at 5,10, 20 minutes,1 and 4 hours
  To assess changes in FEV1 (Forced expiratory volume 1-second) as measured in L.
Change in FEV6 (Forced expiratory volume 6-seconds) | Pre-dose and post-dose at 5, 10, 20 minutes,1 and 4 hours
  To assess changes in FEV6 (Forced expiratory volume 6-seconds) as measured in L.
Change in peak expiratory flow rate (PEFR) | Pre-dose and post-dose at 5, 10, 20 minutes,1 and 4 hours
  To assess changes in PEFR (Peak expiratory flow rate) as measured in L/s.
Change in forced vital capacity (FVC) | Pre-dose and post-dose at 5, 10, 20 minutes,1 and 4 hours
  To assess changes in FVC (Forced vital capacity) as measured by a percentage (%) predicted.
Change in sodium levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in sodium levels as measured in mmol/L.
Change in potassium levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in potassium levels as measured in mmol/L.
Change in chloride levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in chloride levels as measured in mmol/L.
Change in bicarbonate levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in bicarbonate levels as measured in mmol/L.
Change in blood urea nitrogen (BUN) / Urea levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in BUN/Urea levels as measured in mmol/L.
Change in creatinine levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in creatinine levels as measured in umol/L.
Change in total protein levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total protein levels as measured in g/L.
Changes in total albumin levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total albumin levels as measured in g/L.
Change in total ALP levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in ALP levels as measured in U/L.
Change in total ALT levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total ALT levels as measured in U/L.
Change in total AST levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total AST levels as measured in U/L.
Change in total bilirubin levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total bilirubin levels as measured in umol/L.
Change in total indirect bilirubin levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total indirect bilirubin levels as measured in umol/L.
Change in total amylase levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total amylase levels as measured in U/L.
Change in total lipase levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total lipase levels as measured in U/L.
Change in total uric acid levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total uric acid levels as measured in mmol/L.
Change in total creatine kinase (CK) levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total CK levels as measured in U/L.
Change in total calcium levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total calcium levels as measured in mmol/L.
Change in total magnesium levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total magnesium levels as measured in mmol/L.
Change in total lactate dehydrogenase (LDH) levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total LDH levels as measured in U/L.
Change in total immunoglobulin (IgG) levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total IgG levels as measured in g/L.
Change in total immunoglobulin (IgA) levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total IgA levels as measured in g/L.
Changes in total immunoglobulin (IgE) levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total IgE levels as measured in g/L.
Change in total immunoglobulin (IgM) levels as part of standard serum chemistry panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total IgM levels as measured in g/L.
Change in hematocrit as part of standard hematology panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total hematocrit levels as measured by %.
Change in red blood cell (RBC) counts as part of standard hematology panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in total red blood cell (RBC) counts as measured by 10^6/uL.
Change in platelet (PLT) counts as part of standard hematology panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in platelet counts as measured by 10^9/uL.
Change in white blood cell (WBC) counts as part of standard hematology panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in white blood cell (WBC) counts as measured by 10^3/uL.
Change in neutrophil percentage as part of standard hematology panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in neutrophil percentage as measured by %.
Change in lymphocyte percentage as part of standard hematology panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in lymphocyte percentage as measured by %.
Change in eosinophil percentage as part of standard hematology panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in eosinophil percentage as measured by %.
Change in basophil percentage as part of standard hematology panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in basophil percentage as measured by %.
Change in monocyte percentage as part of standard hematology panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in monocyte percentage as measured by %.
Change in clarity as part of a standard urinalysis panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in clarity of the urine sample.
Change in specific gravity as part of a standard urinalysis panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in specific gravity of the urine sample.
Change in pH as part of a standard urinalysis panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in pH of the urine sample.
Change in protein levels as part of a standard urinalysis panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in protein levels of the urine sample.
Change in glucose levels as part of a standard urinalysis panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in glucose levels of the urine sample as measured by a positive or negative result.
Change in ketone levels as part of a standard urinalysis panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in ketone levels of the urine sample as measured by a positive or negative result.
Change in blood levels as part of a standard urinalysis panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in blood levels of the urine sample as measured by a positive or negative result.
Change in nitrite levels as part of a standard urinalysis panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in nitrite levels of the urine sample.
Change in leukocyte esterase levels as part of a standard urinalysis panel. | Screening, day 1, day 2, day 3 and 30 days after dosing.
  To assess changes in leukocyte esterase levels of the urine sample.

SECONDARY OUTCOMES:
PK assessment: Cmax (observed maximum serum concentration taken directly from the individual concentration-time curve) | Pre-dose and post-dose at 5, 10, 20 minutes,1 and 4 hours
  Evaluation of the PK of a single inhaled or IV infusion dose of PRS-060
PK assessment Tmax (Time to reach maximum serum concentration, taken directly from the individual concentration-time curve) | Pre-dose and post-dose at 5, 20 and 40 minutes, 1, 1.5, 2, 3, 4, 8,12,15,18, 36 and 48 hours and at 30 days)
  Evaluation of the PK of a single inhaled or IV infusion dose of PRS-060
PK assessment: t1/2 (Terminal half-life) | Pre-dose and post-dose at 5, 20 and 40 minutes, 1, 1.5, 2, 3, 4, 8,12,15,18, 36 and 48 hours and at 30 days
  Evaluation of the PK of a single inhaled or IV infusion dose of PRS-060
PK assessment: AUC(0-last) (Area under the serum concentration-curve from time zero to the time of last quantifiable analyte concentration) | Pre-dose and post-dose at 5, 20 and 40 minutes, 1, 1.5, 2, 3, 4, 8,12,15,18, 36 and 48 hours and at 30 days
  Evaluation of the PK of a single inhaled or IV infusion dose of PRS-060
PK assessment: AUC (Area under the concentration-time curve in the serum zero (pre-dose) extrapolated to infinite time) | Pre-dose and post-dose at 5, 20 and 40 minutes, 1, 1.5, 2, 3, 4, 8,12,15,18, 36 and 48 hours and at 30 days
  Evaluation of the PK of a single inhaled or IV infusion dose of PRS-060
PK assessment: AUC(0-24) (Area under the plasma concentration-curve) | Pre-dose and post-dose at 5, 20 and 40 minutes, 1, 1.5, 2, 3, 4, 8,12,15,18, 36 and 48 hours and at 30 days
  Evaluation of the PK of a single inhaled or IV infusion dose of PRS-060
PK assessment: Vz/F (Apparent volume of distribution during terminal phase) | Pre-dose and post-dose at 5, 20 and 40 minutes, 1, 1.5, 2, 3, 4, 8,12,15,18, 36 and 48 hours and at 30 days
  Evaluation of the PK of a single inhaled or IV infusion dose of PRS-060
PK assessment: CL/F (Apparent oral clearance estimated as dose divided by AUC) | Pre-dose and post-dose at 5, 20 and 40 minutes, 1, 1.5, 2, 3, 4, 8,12,15,18, 36 and 48 hours and at 30 days
  Evaluation of the PK of a single inhaled or IV infusion dose of PRS-060
PK assessment of urine | Pre-dose and continuously during the following time-intervals: 0-4, 4-8, 8-12, 12-18, 18-24, 24-30, 30-36, 36-42 and 42-48 hours
  Evaluation of PRS-060 levels in the urine after a single inhaled or IV infusion dose of PRS-060

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MBBS PhD, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network Limited, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided